CLINICAL TRIAL: NCT03704740
Title: A Multinational, Comparative Phase III Clinical Trial to Assess the Efficacy (Immunogenicity) and Safety of NBP607-QIV (0.5 mL) (Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine) in Children Aged 6 to 35 Months
Brief Title: Immunogenicity and Safety of NBP607-QIV Compared to Agrippal in Children Aged 6 to 35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607-QIV_005
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP607-QIV (Experimental): One or two doses of 0.5mL of NBP607-QIV by intramuscular injection
  Interventions: Biological: NBP607-QIV
- Agrippal (Active Comparator): One or two doses of 0.25mL of Agrippal by intramuscular injection
  Interventions: Biological: Agrippal

INTERVENTIONS:
Biological: NBP607-QIV — Purified inactivated influenza virus surface antigens of four strains (quadrivalent)
  Arms: NBP607-QIV
Biological: Agrippal — Influenza virus surface antigens of three strains (trivalent)
  Arms: Agrippal

SUMMARY:
This study assesses immunogenicity and safety of NBP607-QIV to Agrippal which are indicated for active immunization for the prevention of influenza disease. Total of 675 subjects or above (450 subjects for NBP607-QIV arm and 225 subjects for Agrippal arm) of 6 to 35 months of age are enrolled, and each subject is administered with single or two doses of vaccines depending on previous vaccination history.

DETAILED DESCRIPTION:
This is a multi-national, multi-center, randomized, double blinded, parallel-group study to assess the immunogenicity and safety of NBP607-QIV compared to Agrippal which are indicated for active immunization for the the prevention of influenza disease. Total of 675 subjects or above (450 subjects for NBP607-QIV arm and 225 subjects for Agrippal arm) of 6 to 35 months of age are enrolled. Each subject is administered with single or two doses of vaccines depending on previous vaccination history, and randomly assigned in 2:1 ratio.

Stratified randomization for trial site and age strata is used to achieve the balance of treatment assignment.

Total of three or five visits are scheduled depeding on dosing schedule. For subjects assigned to single-dose vaccination schedule, blood sampling is conducted for immunogenicity assessment before and 4 weeks after single vaccination at Visit 1 and 3 respectively. Safety is monitored 3 days, 4 weeks after vaccination through Visit 2* and 3 (* telephone contact). For subjects assigned to two-dose vaccination schedule, blood sampling is conducted before first vaccination and 4 weeks after second vaccination at Visit 1 and Visit 5 respectively. Safety is monitored 3 days, 4 weeks after each vaccination through Visit 2*, 3, 4*, and 5 (* telephone contact)

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 35 months
* Those who were normal gestational age at birth (for children aged 6 months to <1 year)
* Those who have provided written informed consent to study participation and compliance with study instructions after being informed of and understand details of the study

Exclusion Criteria:

* Those with any immunodeficiency disease or malignancy
* Those with hypersensitivity to vaccination
* Those who are contraindicated for intramuscular injection due to thrombocytopenia or other coagulopathy
* Those with history of treatment with any of immunosuppressants or immunoregulators within 12 weeks prior to screening
* Those with history of receiving blood product or treatment with immunoglobulin within 24 weeks prior to screening
* Those with history of influenza vaccination within 24 weeks prior to screening
* Those with any severe chronic conditions that interfere with study participation

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 676 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Post-vaccination GMT(Geometric Mean Titer) by HI(Hemagglutination-inhibition) assay for the common strains (A/H1N1, A/H3N2, and B/Victoria) | 4 weeks after last IP(Investigational Product) vaccination
  Post-vaccination GMT will be adjusted for pre-vaccination titer
Seroconversion rate by HI assay for the common strains (A/H1N1, A/H3N2, and B/Victoria) | 4 weeks after last IP(Investigational Product) vaccination
  Seroconversion rate is defined as the proportion of subjects who meet either of the following criteria:
  1. Post-vaccination HI titer of ≥1:40 for subjects with pre-vaccination HI titer of <1:10
  2. Four-fold increase in post-vaccination HI titer for subjects with pre-vaccination HI titer of ≥1:10
Seroconversion rate by HI assay for the exclusive strain (B/Yamagata) | 4 weeks after last IP(Investigational Product) vaccination
  Seroconversion rate is defined as the proportion of subjects who meet either of the following criteria:
  1. Post-vaccination HI titer of ≥1:40 for subjects with pre-vaccination HI titer of <1:10
  2. Four-fold increase in post-vaccination HI titer for subjects with pre-vaccination HI titer of ≥1:10
GMR(Geometric mean ratio) by HI assay for the exclusive strain (B/Yamagata) | 4 weeks after last IP(Investigational Product) vaccination
  The fold-rise of the geometric mean HI titer from pre- to post-vaccination

SECONDARY OUTCOMES:
Seroprotection rate by HI assay for all strains | 4 weeks after last IP(Investigational Product) vaccination
  Seroprotection rate is defined as the proportion of subjects whose post-vaccination HI titer increased to ≥1:40
CHMP(Committee for Medicinal Products for Human Use) criteria assessment for the common strains (A/H1N1, A/H3N2, and B/Victoria) | 4 weeks after last IP(Investigational Product) vaccination
  CHMP criteria for seroconversion rate, GMR(Geometric Mean Ratio) will be assessed
Consistency of immunogenicity among countries | 4 weeks after last IP(Investigational Product) vaccination
  Post-vaccination GMT and seroconversion rate for the common strains (A/H1N1, A/H3N2, and B/Victoria), and CHMP criteria for seroconversion rate and GMR for the exclusive strain (B/Yamagata) will be assessed
Percentage of participants with Adverse Events(AEs) | 7 days for Solicited AE and 4 weeks for Unsolicited AE, SAE after last IP(Investigational Product) vaccination
  Incidence rate of Solicited AE, unsolicited AE, SAE(Serious Adverse Event) will be assessed
Vital sign | 4 weeks after last IP(Investigational Product) vaccination
  Body temperature will be assessed
Height | 4 weeks after last IP(Investigational Product) vaccination
  Height in centimeters will be assessed
Weight | 4 weeks after last IP(Investigational Product) vaccination
  Weight in kilograms will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kyung Kim, MD, Study Chair — Korea University
Locations (1):
- SK Bioscience, Gyeonggi-do, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No